CLINICAL TRIAL: NCT01195363
Title: A Randomized, Double-Blind, Placebo Controlled Study Of Quetiapine SR (QTP) As Adjunctive Treatment In Mixed States (MS) Of Bipolar Disorder
Brief Title: Quetiapine Sr as Adjunctive Treatment In Mixed States of Bipolar Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Charles L. Bowden, MD, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC20070253H
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder, mania, depression
MeSH Terms: conditions — Bipolar Disorder; Mania; Depression | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- quetiapine SR (Active Comparator): quetiapine SR, 200-600mg, po, qd
  Interventions: Drug: quetiapine SR
- quetiapine sr Placebo (Placebo Comparator): quetiapine SR placebo, 200-600mg, po qd
  Interventions: Drug: quetiapine sr placebo

INTERVENTIONS:
Drug: quetiapine SR — quetiapine SR, dose range 200-600mg, each night QHS for 6mos
  Other Names: Seroquel SR
  Arms: quetiapine SR
Drug: quetiapine sr placebo — quetiapine sr placebo, dose range 200-600mg, each night QHS for 6mos
  Arms: quetiapine sr Placebo

SUMMARY:
To assess the acute and long-term bimodal efficacy of QTP, as an adjunct to ongoing treatment with lithium (Li) or divalproex (DIV) or lamotrigine (LAM) or any combination of the three thereof, in a group of patients with an index episode of a mixed state in BD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* Age 18 years and older
* Patients on:

  * Li at a stable dose for 4 weeks or longer, and a serum level at screening of 0.5 mEq/l OR
  * DIV dose for 4 weeks or longer, and a serum level at screening of 45 g/ml OR
  * LAM (dosage/day ≥100mg) at a stable dose for 4 weeks or longer OR
  * Any combination 3a, 3b, or 3c
* Patients meeting DSM-IV TR diagnosis of bipolar disorder, I or II, as assessed using the MINI, (Sheehan et al., 1998) PLUS any ONE of criteria 5 or 6 or 7
* Patients meeting DSM-IV TR diagnostic criteria for a mixed manic episode with Young Mania Rating Scale (YMRS) score>/=14 and Montgomery Asberg Depression Rating Scale (MADRS) score>/=14
* Patients meeting the criteria for a manic/hypomanic episode for at least 2 days with the simultaneous presence of Young Mania Rating Scale (YMRS) score>/=14 PLUS Montgomery Asberg Depression Rating Scale (MADRS) score>/=14 ;
* Patients meeting DSM-IV TR diagnostic criteria for a major depressive episode with the simultaneous presence of MADRS score>/=14 PLUS meeting the criteria for a manic/hypomanic episode for at least 2 days with the simultaneous presence of Young Mania Rating Scale (YMRS) score>/=14

Exclusion Criteria:

* Patients with a current Axis I diagnosis of schizophrenia, schizophreniform disorder, schizotypal disorder, bipolar disorder with psychotic subtype, drug induced mania or AIDS induced mania
* Women with a positive pregnancy test or who are lactating
* Women of child-bearing potential who are not practicing a clinically accepted method of contraception
* Patients with general medical conditions that contraindicate psychoactive medications or uncontrolled medical disorder or central nervous system diseases.
* Patients whose clinical status requires inpatient or day hospital treatment
* History of severe side effects associated with therapeutic doses of Li, DIV, LAM
* Alcohol or drug dependent at time of enrollment
* Suicidal at time of enrollment.
* Current or previous exposure to QTP

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-04; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bowden, MD, Principal Investigator — University of Texas
Locations (1):
- The University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in our University, Center for Healthcare Services, and by televison ads between Oct 2007 and January 2011.
Pre-assignment Details: Patients screened over a 7 day period.
Groups:
- Quetiapine SR, 200-600mg , po, QD: mood stabilizer plus active quetiapine SR
- Quetiapine sr Placebo 200-600mg, po, qd: mood stabilizer plus quetiapine SR placebo
Period: Overall Study
Arm/Group | Quetiapine SR, 200-600mg , po, QD | Quetiapine sr Placebo 200-600mg, po, qd
Started | 15 | 13
Completed | 4 | 4
Not Completed | 11 | 9
Not completed — Lost to Follow-up | 7 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Lack of Efficacy | 0 | 4
Not completed — incarceration | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Quetiapine SR: mood stabilizer plus active quetiapine sr
- Quetiapine SR Placebo: mood stabilizer plus quetiapine SR placebo
- Total: Total of all reporting groups
Arm/Group | Active Quetiapine SR | Quetiapine SR Placebo | Total
Number analyzed (Participants) | 15 | 13 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 13 | 28
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.5 (10.1) | 32.1 (9.8) | 34 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 7 | 2 | 9
Region of Enrollment [Number; unit: participants]
  United States | 15 | 13 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Whose Mood Improved According to MADRS and YMRS Scale Scores.
Description: The primary outcome measure was assessed by 50% reduction in: 1. depression scores on the Montgomery Asberg Depression Rating Scale (MADRS), which ranges from 0 indicating no symptoms to 60 indicating most symptoms 2. mania scores on the Young Mania Rating Scale (YMRS), which ranges from 0 indicating no symptoms to 60 indicating most symptoms.
Time Frame: Baseline visit to week 24
Population: Per Protocol
Measure: Number; unit: participants
Groups:
- Active Quetiapine S.R., 200-600mg, po, qd: Atypical antipsychotic quetiapine S.R. plus mood stabilizer
- Placebo Quetiapine S.R. 200-600mg, po, qd: mood stabilizer plus quetiapine S.R. placebo
Arm/Group | Active Quetiapine S.R., 200-600mg, po, qd | Placebo Quetiapine S.R. 200-600mg, po, qd
Number analyzed (Participants) | 15 | 13
participants
  MADRS | 4 | 4
  YMRS | 4 | 4

ADVERSE EVENTS:
Time Frame: 10/30/2007 - 6/1/2011, 2 yrs 8 mos.
Groups:
- Mood Stabilizer Plus Quetiapine SR: mood stabilizer plus active quetiapine SR
- Mood Stabilizer Plus Quetiapine sr Placebo: mood stabilizer plus quetiapine SR placebo
Arm/Group | Mood Stabilizer Plus Quetiapine SR | Mood Stabilizer Plus Quetiapine sr Placebo
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 10/15 | 7/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mood Stabilizer Plus Quetiapine SR (N=15) | Mood Stabilizer Plus Quetiapine sr Placebo (N=13)
dry mouth (General disorders) | 4 (4) | 2 (2)
joint pain (General disorders) | 2 (2) | 0 (0)
drowsiness/sedation (Investigations) | 7 (7) | 3 (3)
interrupted sleep (Investigations) | 2 (2) | 0 (0)
muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
headache (General disorders) | 1 (1) | 2 (2)
increased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Overall limitations were screen failures and lost to follow-ups which led to not reaching recruitment goals.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No